CLINICAL TRIAL: NCT00939354
Title: Asthma in the Elderly: The Role of Exhaled Nitric Oxide Measurements
Status: Completed | Type: Observational
Sponsor: Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C. (Other)
Responsible Party: Principal Investigator, Michele Columbo, M.D., Co-Investigator, Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C.
Other Study IDs: F/N-R09-2839B
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Asthma
Keywords: Asthma in subjects over the age of 65
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will investigate the importance of exhaled nitric oxide measurements in subjects with asthma age 65 and older. This group of patients has been ignored in most previous asthma studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with asthma over the age of 65 followed in our practice, non-smokers and able to give informed consent to participate in the study

Exclusion Criteria:

* Smokers, subjects of diminished mental capacity

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Subjects with asthma over the age of 65 who are currently followed in our practice
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Exhaled Nitric Oxide (FENO) levels and their changes with time | One year

SECONDARY OUTCOMES:
Correlations of FENO with subjects' demographics, comorbidities, treatment, symptoms, or spiromentric values | One year

CONTACTS AND LOCATIONS:
Overall Officials: Albert S Rohr, M.D., Principal Investigator — Rohr and Columbo Associates